CLINICAL TRIAL: NCT00017719
Title: Randomized Trial of Protease Inhibitor-Including vs. Protease Inhibitor-Sparing Regimens for Women Who Initiate Therapy of HIV Infection During Pregnancy
Brief Title: Combination Treatment With and Without Protease Inhibitors for Women Who Begin Therapy for HIV Infection During Pregnancy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: P1022; 10192 (Registry Identifier: DAIDS ES); ACTG P1022; PACTG P1022
Record Dates: First submitted 2001-06-08; First posted 2001-08-31 (Estimated); Last update posted 2021-11-01 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections; Pregnancy
Keywords: Pregnancy Complications, Infectious; HIV Protease Inhibitors; Reverse Transcriptase Inhibitors; Anti-HIV Agents; Viral Load; Combivir; Treatment Naive
MeSH Terms: conditions — HIV Infections; Pregnancy Complications, Infectious | interventions — Lamivudine; lamivudine, zidovudine drug combination; Nelfinavir; Nevirapine; Zidovudine

INTERVENTIONS:
Drug: Lamivudine
Drug: Lamivudine/Zidovudine
Drug: Nelfinavir mesylate
Drug: Nevirapine
Drug: Zidovudine

SUMMARY:
The best anti-HIV treatment regimen for pregnant women is not known. Protease inhibitors (PIs) are often used, but they have side effects that may be harmful for pregnant women. It is not known if treatment regimens that do not include PIs are as effective in pregnant women as those that include PIs. This trial will compare two anti-HIV treatment plans, one with and one without PIs, in women who start HIV treatment during pregnancy. The study will evaluate the effects of the anti-HIV drugs on the developing infant and prevention of mother-to-child HIV transmission during pregnancy.

DETAILED DESCRIPTION:
The optimal treatment strategy for women who initiate antiretroviral therapy during pregnancy is not known. Although PI-based antiretroviral regimens are prescribed with increasing frequency among pregnant women, the efficacy and safety of this approach is unknown. Pregnant women are at increased risk for glucose intolerance and insulin resistance; PIs are associated with glucose intolerance. Physiologic differences between pregnant women and nonpregnant adults may alter the pharmacokinetics of antiretroviral regimens. Fetal safety considerations and effects on perinatal HIV transmission must also be considered when selecting an antiretroviral regimen for pregnant women. This trial will compare PI-based and PI-sparing antiretroviral regimens for women initiating antiretroviral therapy in pregnancy.

Women will be stratified on the basis of viral load (50,000 or less copies/ml or greater than 50,000 copies/ml) and gestational age at entry (20 or less weeks or greater than 20 weeks) and then randomized to one of two treatment groups. Group A will receive the PI nelfinavir (NFV) with zidovudine (ZDV) and lamivudine (d4T); Group B will receive nevirapine (NVP) with ZDV and d4T. Women will have clinic visits for physical and obstetrical examinations at 2, 4, 6, and 8 weeks after entry and then every 4 weeks until delivery. After delivery, infants in both groups may receive ZDV until they are 6 weeks old. Infants are evaluated for safety and to test the infant's blood for HIV-1 at birth and at Weeks 2, 8, 16, and 24.

Women will continue on assigned antiretroviral therapy postpartum and will have 11 postpartum clinic visits over a period of 2 years. Blood samples from women will be evaluated for safety and for virologic, pharmacokinetic, and metabolic studies. The first 12 women randomized to Group A will undergo a 4-hour pharmacokinetic profile at 32 to 36 weeks gestation and at 8 weeks postpartum to determine the timing of the nelfinavir trough. The first 20 women randomized to Group B will undergo an 8-hour pharmacokinetic profile at either 16 to 24 weeks or 32 to 36 weeks gestation and then again at 8 weeks postpartum to characterize pharmacokinetics of nevirapine at steady state in pregnancy and in the postpartum period.

ELIGIBILITY:
Inclusion Criteria:

* HIV infected
* 10 to 30 weeks pregnant
* Plan to continue pregnancy
* CD4 count less than 250 cells/mm3 within 30 days of study entry
* HIV RNA load greater than 1,000 copies/ml within 30 days of study entry
* Antiretroviral naive (except ZDV for 8 weeks or less, including prior pregnancy)
* Willing to follow study requirements and plan to continue receiving anti-HIV treatment for at least 2 years after delivery
* Understand that NFV will not be supplied by the study (except for the first 12 women in Group A)
* Understand the study drug NVP will not be supplied after 1 year following delivery and is reasonably certain that she can obtain NVP by prescription for the second year of the study
* Access to a participating site
* Willing to have infant followed until 24 weeks old
* Parent or guardian willing to provide informed consent, if applicable

Exclusion Criteria:

* Alcohol or drug abuse
* Chemotherapy for an active cancer
* Require certain medications
* AIDS-related opportunistic infection and/or serious bacterial infection or unstable or serious medical condition within 14 days of study entry
* Chronic malabsorption or diarrhea
* Diabetes, unless it only occurs during pregnancy
* Major fetal problem or abnormality
* Abnormal amniotic fluid volume
* Plan to breastfeed
* Acute hepatitis within 90 days of study entry
* Skin problems such as psoriasis or eczema that require systemic treatment
* Any serious disease that, in the opinion of the study official, would compromise study participation

Min Age: 14 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 440
Dates: Start 2002-05; Study Completion 2006-03 (Actual)

PRIMARY OUTCOMES:
Proportion of women in each treatment group who continue on original therapy with virologic suppression to less than 500 copies/ml at 34 weeks gestation (or the last viral load determination prior to delivery)
proportion of women in each treatment group who continue on original therapy with virologic suppression to less than 500 copies/ml at 48 weeks postpartum

SECONDARY OUTCOMES:
Proportion of women in each treatment group who continue on original therapy with virologic suppression to less than 50 copies/ml at 34 weeks gestation (or the last viral load determination prior to delivery)
proportion of women in each treatment group who continue on original therapy with virologic suppression to less than 50 copies/ml at 48 weeks postpartum, and to less than 500 and 50 copies/ml at 104 weeks postpartum
study treatment adherence and health status by self-report, correlated with predose nelfinavir or nevirapine level at 34 weeks gestation and 8 weeks postpartum
difference between postpartum and pregnancy 12-hour area under the concentration curve (AUC) for nevirapine
time of trough levels in relation to the morning dose of nevirapine and nelfinavir at 34 weeks gestation and 8 weeks postpartum and correlation of trough levels with viral load
incidence of HIV viral resistance by genotype among women in each treatment group at the time of virologic failure
incidence of abnormal glucose tolerance, gestational diabetes, and abnormal lactate levels during pregnancy in each treatment group
incidence of impaired glucose tolerance, diabetes, hyperinsulinemia, and elevated cholesterol and triglycerides at 8 weeks postpartum in each treatment group
incidence of anemia, hypoglycemia, and abnormal liver function studies among infants born to women in each treatment group
incidence of prematurity (less than 37 weeks), extreme prematurity (less than 32 weeks), low birth weight (less than 2.5 kg), and very low birth weight (less than 1.5 kg) among infants born to women in each treatment group
perinatal HIV transmission among infants born to women in each treatment group

CONTACTS AND LOCATIONS:
Overall Officials: Jane Hitti, MD, MPH, Study Chair — Department of Obstetrics/Gynecology, University of Washington Medical Center
Locations (49):
- United States (44):
  - Usc La Nichd Crs, Los Angeles, California
  - UCSD Mother-Child-Adolescent Program CRS, San Diego, California
  - UCSF Pediatric AIDS CRS, San Francisco, California
  - Harbor - UCLA Med. Ctr. - Dept. of Peds., Div. of Infectious Diseases, Torrance, California
  - Yale Univ. School of Medicine - Dept. of Peds., Div. of Infectious Disease, New Haven, Connecticut
  - Howard Univ. Washington DC NICHD CRS, Washington D.C., District of Columbia
  - Univ. of Miami Miller School of Medicine - Jackson Memorial Hosp., Miami, Florida
  - Univ. of Miami Ped. Perinatal HIV/AIDS CRS, Miami, Florida
  - Med. College of Georgia School of Medicine, Dept. of Peds., Div. of Infectious Diseases, Augusta, Georgia
  - Columbus Regional HealthCare System, The Med. Ctr., Columbus, Georgia
  - Mt. Sinai Hosp. Med. Ctr. - Chicago, Womens & Childrens HIV Program, Chicago, Illinois
  - Univ. of Chicago - Dept. of Peds., Div. of Infectious Disease, Chicago, Illinois
  - Tulane Univ. Health Science Ctr., Tulane Univ. Hosp. & Clinic, New Orleans, Louisiana
  - Tulane/LSU Maternal/Child CRS, New Orleans, Louisiana
  - Johns Hopkins Hosp. & Health System - Dept. of Peds., Div. of Infectious Diseases, Baltimore, Maryland
  - Univ. of Maryland Med. Ctr., Div. of Ped. Immunology & Rheumatology, Baltimore, Maryland
  - HMS - Children's Hosp. Boston, Div. of Infectious Diseases, Boston, Massachusetts
  - BMC, Div. of Ped Infectious Diseases, Boston, Massachusetts
  - Brigham and Women's Hosp., Div. of Infectious Disease, Boston, Massachusetts
  - Baystate Health, Baystate Med. Ctr., Springfield, Massachusetts
  - WNE Maternal Pediatric Adolescent AIDS CRS, Worcester, Massachusetts
  - Children's Hospital of Michigan NICHD CRS, Detroit, Michigan
  - Univ. of Mississippi Med. Ctr Children's Hosp., Jackson, Michigan
  - Rutgers - New Jersey Medical School CRS, Newark, New Jersey
  - Nyu Ny Nichd Crs, New York, New York
  - Columbia IMPAACT CRS, New York, New York
  - Strong Memorial Hospital Rochester NY NICHD CRS, Rochester, New York
  - SUNY Stony Brook NICHD CRS, Stony Brook, New York
  - SUNY Upstate Med. Univ., Dept. of Peds., Syracuse, New York
  - Bronx-Lebanon Hosp. IMPAACT CRS, The Bronx, New York
  - Montefiore Med. Ctr. - AECOM, The Bronx, New York
  - DUMC Ped. CRS, Durham, North Carolina
  - Univ. of Cincinnati CRS, Cincinnati, Ohio
  - Case CRS, Cleveland, Ohio
  - MetroHealth CRS, Cleveland, Ohio
  - Oregon Health & Science Univ. - Dept. of Peds., Div. of Infectious Disease, Portland, Oregon
  - Regional Med. Ctr. at Memphis, Memphis, Tennessee
  - St. Jude/UTHSC CRS, Memphis, Tennessee
  - Vanderbilt Univ. Med. Ctr., Div. of Ped. Infectious Diseases, Nashville, Tennessee
  - Texas Children's Hosp. CRS, Houston, Texas
  - Univ. of Washington NICHD CRS, Seattle, Washington
  - UW Medicine - Harborview Med. Ctr., Northwest Family Ctr., Seattle, Washington
  - UW School of Medicine - CHRMC, Seattle, Washington
  - Seattle Children's Hospital CRS, Seattle, Washington
- Brazil (3):
  - SOM Federal University Minas Gerais Brazil NICHD CRS, Belo Horizonte, Minas Gerais
  - Hosp. dos Servidores Rio de Janeiro NICHD CRS, Rio de Janeiro
  - Hosp. dos Servidores do Estado CRS, Rio de Janeiro
- San Juan City Hosp. PR NICHD CRS, San Juan, Puerto Rico
- Princess Margaret Hosp. Bahamas NICHD CRS, Nassau, The Bahamas

REFERENCES:
- [Background] Loutfy MR, Walmsley SL. Treatment of HIV infection in pregnant women: antiretroviral management options. Drugs. 2004;64(5):471-88. doi: 10.2165/00003495-200464050-00002. PMID 14977385
- [Background] Moodley J, Moodley D. Management of human immunodeficiency virus infection in pregnancy. Best Pract Res Clin Obstet Gynaecol. 2005 Apr;19(2):169-83. doi: 10.1016/j.bpobgyn.2004.10.007. Epub 2004 Dec 15. PMID 15778108
- [Result] Hitti J, Frenkel LM, Stek AM, Nachman SA, Baker D, Gonzalez-Garcia A, Provisor A, Thorpe EM, Paul ME, Foca M, Gandia J, Huang S, Wei LJ, Stevens LM, Watts DH, McNamara J; PACTG 1022 Study Team. Maternal toxicity with continuous nevirapine in pregnancy: results from PACTG 1022. J Acquir Immune Defic Syndr. 2004 Jul 1;36(3):772-6. doi: 10.1097/00126334-200407010-00002. PMID 15213559
- [Result] Capparelli EV, Aweeka F, Hitti J, Stek A, Hu C, Burchett SK, Best B, Smith E, Read JS, Watts H, Nachman S, Thorpe EM Jr, Spector SA, Jimenez E, Shearer WT, Foca M, Mirochnick M; PACTG 1026S Study Team; PACTG P1022 Study Team. Chronic administration of nevirapine during pregnancy: impact of pregnancy on pharmacokinetics. HIV Med. 2008 Apr;9(4):214-20. doi: 10.1111/j.1468-1293.2008.00553.x. PMID 18366444